CLINICAL TRIAL: NCT02628561
Title: Transcranial Direct Current Stimulation Associate to Constraint Induced Movement Therapy Over Premotor Cortex in Severe Stroke
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Suellen Marinho Andrade, PhD, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: tdcstroke
Record Dates: First submitted 2015-12-04; First posted 2015-12-11 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Stroke; Cerebrovascular Disorders; Cerebral Infarction
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Cerebral Infarction | interventions — Transcranial Direct Current Stimulation; Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active tdcs/M1 (Active Comparator): Anodal tDCS on primary motor cortex and CIMT (constraint induced movement therapy)
  Interventions: Device: Transcranial direct current stimulation; Behavioral: Constraint-Induced Movement Therapy
- Active tdcs/Premotor (Experimental): Anodal tDCS on premotor cortex and CIMT (constraint induced movement therapy)
  Interventions: Device: Transcranial direct current stimulation; Behavioral: Constraint-Induced Movement Therapy
- Sham tdcs (Sham Comparator): Sham tDCS and CIMT (constraint induced movement therapy)
  Interventions: Device: Transcranial direct current stimulation; Behavioral: Constraint-Induced Movement Therapy

INTERVENTIONS:
Device: Transcranial direct current stimulation
Behavioral: Constraint-Induced Movement Therapy

SUMMARY:
The purpose is to compare the effects of tDCS and constraint induced movement therapy (CIMT) in the premotor cortex vs. primary motor cortex in severely subacute stroke survivors.

DETAILED DESCRIPTION:
Stroke survivors experience one or more movement-related impairments and activity limitations. In this sense, the premotor cortex (PMC) can be considered as an alternative locus for post-stroke rehabilitation. In relation to physical rehabilitation protocols, associate to neuromodulation, the investigators have chosen a standardized physical therapy protocol for this study, the Constraint Induced Movement Therapy (CIMT), which presents evidence of good therapeutic results. The investigators hypothesized that applying tDCS and CIMT over the PMC promotes motor restoration in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Diagnosis of unilateral, non-recurring, subacute stroke
* Participants also had to be able, by using any method of pinch, to grasp a washcloth from a table top, lift it up a few inches, and release it.

Exclusion Criteria:

* Patients with difficulty to follow the procedures or understand the instructions; cognitive deficits
* tDCS criteria:

  * use of modulators of the Central Nervous System drugs
  * patients with implanted metallic or electronic devices
  * pacemaker
  * seizures
  * pregnancy
  * any other condition that might limit or interfere in the sensorimotor system

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Functional Independence measured by Barthel Index | Change for functional independence at baseline and week 2

SECONDARY OUTCOMES:
Spasticity (Modified Ashworth Scale) | Baseline and Week 2
Muscle strength (Medical Research Council Scale) | Baseline and Week 2

CONTACTS AND LOCATIONS:
Locations (1):
- Suellen Andrade, João Pessoa, Paraíba, Brazil